CLINICAL TRIAL: NCT06133296
Title: Comparison of Anxiety, Pain, and Quality of Life in Individuals With Moderate Malocclusion Between Conventional Fixed Treatment and Invisalign: a Randomized Clinical Trial
Brief Title: Anxiety, Pain, and Quality of Life in Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Murat Tunca, PhD, DDS, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021/02-08
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Malocclusion; Pain; Anxiety; Quality of Life
Keywords: clear aligner; Anxiety; Pain; Quality of Life
MeSH Terms: conditions — Malocclusion; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Conventional fixed treatment) (Active Comparator): Roth brackets (.018; Gemini Roth System, 3M Unitek, USA) were used for the fixed orthodontic attachment. Tooth surfaces were etched with 35% gel phosphoric acid for 30 seconds and then washed with water for 15 seconds. A primer was applied to the etching surface with the manufacturer's applicator. After an adhesive was applied to the bases of the brackets, the brackets were placed in their appropriate positions. Afterward, LED was irradiated for 20 seconds and 5 seconds for each surface. For leveling after bonding, .012 nickel titanium archwires (3M Unitek Monrovia, CA, USA) were tied with an elastic ligature.
  Interventions: Other: Conventional fixed treatment
- Group B (Clear aligner treatment) (Active Comparator): Clear aligners were ordered after the recordings were evaluated in the Clincheck program, and the final treatment plan was created. After the clear aligners came from the manufacturer (Align Technology, Santa Clara, CA), the compatibility of the guide aligner with each patient's mouth was checked for attachments. The enamel surfaces on which the attachments will be applied were etching with the same method as in Group A. After an adhesive was condensed into the attachment spaces inside the guide plate, the guide aligner was placed in the correct position in the mouth, and each attachment was applied from the buccal surface with an LED light device for 20 seconds. After the guide plate was removed, the composite residues around the attachments were cleaned, and the first treatment aligner was applied. The individuals were informed that they should use their clear aligner continuously, except during meals, and replace them after 10 days.
  Interventions: Other: Clear aligner treatment

INTERVENTIONS:
Other: Conventional fixed treatment — Roth brackets (.018; Gemini Roth System, 3M Unitek, USA) were used for the fixed orthodontic attachment
  Arms: Group A (Conventional fixed treatment)
Other: Clear aligner treatment — After the clear aligners came from the manufacturer (Align Technology, Santa Clara, CA), the compatibility of the guide aligner with each patient's mouth was checked for attachments
  Arms: Group B (Clear aligner treatment)

SUMMARY:
This study was evaluated anxiety, pain, and oral health-related quality of life in individuals treated with conventional fixed appliances (Group A) and clear aligners (Group B) for moderate malocclusion during the initial phase of orthodontic treatment

DETAILED DESCRIPTION:
Clear aligner treatment is becoming increasingly popular among orthodontic treatment option. With this treatment method, which was introduced the literature at the beginning of the 20th century, approximately four million individuals in 2019 and over twelve million individuals have already been treated today. In addition, the number of commercial companies worldwide producing transparent plaque has reached twenty-seven, indicating that these figures will increase rapidly. Although there are debates about the effectiveness of the treatment, the increase in living standards and the improvement of the quality of life of individuals relative to conventional fixed orthodontic treatment have increased interest in clear aligner treatment.

The World Health Organization has multidimensional definitions of the concepts of "quality of life" and "health," and their common point is that they emphasize the importance of the psychological and social status of individuals in recent years. Quality of life is affected by dentofacial problems caused by malocclusions, as well as the psychosocial state of individuals during orthodontic treatment. Oral health-related quality of life was defined as "the absence of physical and psychological problems in terms of oral health and self-confidence associated with the maxillofacial region," and the importance of self-confidence and psychosocial status that could affect quality of life was emphasized. The presence of pain and anxiety before and at the beginning of orthodontic treatment are among the factors affecting oral health-related quality of life.

Pain is an emotional state frequently encountered by individuals undergoing orthodontic treatment, leading to cooperation problems and even causing them to give up treatment. In studies comparing the pain levels of individuals treated with conventional fixed orthodontic appliances and clear aligners, individuals treated with clear aligners felt less pain in the first few days, but there was no significant difference in pain levels in later periods of treatment.

The importance of malocclusion type and arc length disperancy has been emphasized in studies comparing conventional fixed therapy and clear plating therapy in terms of pain and quality of life. Considering that the concepts of anxiety, pain, and quality of life are interrelated by each other, there are limited studies in which both treatment methods are evaluated in terms of these factors in a particular malocclusion. The current study aims to compare anxiety and pain values observed in the initial phase of orthodontic treatment and oral health-related quality of life among individuals with moderate malocclusion treated with conventional fixed orthodontic appliances and clear aligners. Our null hypothesis (H0) is that there is no difference in anxiety, pain, or oral health-related quality of life between individuals treated with conventional fixed orthodontic appliances and clear aligners.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who had not received orthodontic treatment before,
* Angle class I malocclusion,
* 4-6 mm arc length disperancy in both dental arches,
* Permanent dentition period,
* Missing or impacted teeth,
* No smoker,
* No alcohol drinker.

Exclusion Criteria:

* Individuals who underwent extraction fixed orthodontic treatment,
* Radiologically observed alveolar bone loss,
* Missing or impacted teeth,
* systemic disease,
* Using of drugs or analgesics.

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
VAS | 0 hour, 2 hours, 6 hours, 1st day, 3rd day, 7th day, 14th day, 21st day.
  Visual Analogue Scale (VAS) was used to measure the individuals' pain levels. VAS is a scale that ranges pain severity from 0 to 10. (0= no pain, 10= severe pain)
OHIP-14 | Baseline, 10th day, 20th day
  The Oral Health Impact Profile-14 (OHIP-14) questionnaires were used to measure quality of life in our study. The OHIP-14 questionnaire consists of seven domains and 14 questions, including those related to functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, and disability. The individuals were asked to answer each question as follows: 0: never, 1: very little, 2: sometimes, 3: quite often, and 4: often. After the results were collected separately for each of the seven subgroups, they were added together to calculate the actual results. High scores obtained on the OHIP-14 questionnaire indicate that quality of life was adversely affected.
OHRQoL-UK | Baseline, 10th day, 20th day
  The Oral Health-Related Quality of Life-United Kingdom (OHRQoL-UK) questionnaires were used to measure quality of life in our study. In the OHRQoL-UK questionnaire, 16 questions were asked in four categories: symptom (two questions), physical condition (five questions), psychological condition (five questions), and social situation (four questions).Answers scored according to the Likert scale were given 1 point for very bad influence, 2 for bad influence, 3 for no effect, 4 for good effect, and 5 for very good effect. The scores ranged from 16 to 80. A high score indicates a good quality of life for oral and dental health, whereas a low score indicates a poor quality of life for oral and dental health.

SECONDARY OUTCOMES:
Anxiety | Before treatment, baseline, 10th day, and 20th day.
  The Spielberger State and Trait Anxiety Inventory (STAI) survey was applied. It includes 40 questions that measure state anxiety (STAI-S, 20) and trait anxiety (STAI-T, 20). The answer categories for the questions varied according to the nature of the problem (e.g., 1: No, 2: slightly, 3: multiple, and 4: always) in the form of a four-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Tunca, PhD, DDS, Principal Investigator — Yuzuncu Yil University; Yesim Kaya, PhD, DDS, Study Chair — Ankara Yildirim Beyazıt University; Yasemin Tunca, PhD, DDS, Study Chair — Yuzuncu Yil University; Siddik Keskin, PhD, DDS, Study Chair — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfawal AMH, Burhan AS, Mahmoud G, Ajaj MA, Nawaya FR, Hanafi I. The impact of non-extraction orthodontic treatment on oral health-related quality of life: clear aligners versus fixed appliances-a randomized controlled trial. Eur J Orthod. 2022 Dec 1;44(6):595-602. doi: 10.1093/ejo/cjac012. PMID 35395075
- [Background] Flores-Mir C, Brandelli J, Pacheco-Pereira C. Patient satisfaction and quality of life status after 2 treatment modalities: Invisalign and conventional fixed appliances. Am J Orthod Dentofacial Orthop. 2018 Nov;154(5):639-644. doi: 10.1016/j.ajodo.2018.01.013. PMID 30384934
- [Derived] Tunca Y, Kaya Y, Tunca M, Keskin S. Comparison of anxiety, pain, and quality of life in individuals with mild or moderate malocclusion between conventional fixed orthodontic treatment versus Invisalign: a randomised clinical trial. BMC Oral Health. 2024 May 17;24(1):576. doi: 10.1186/s12903-024-04335-1. PMID 38760747